CLINICAL TRIAL: NCT02977897
Title: Fecal Calprotectin Levels in Mycophenolate Mofetil Induced Diarrhea and Treatment With Octreotide
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-5998
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Diarrhea; Immunosuppression
Keywords: Diarrhea; Immunosuppression; Post-transplantation; Octreotide; Mycophenolate Mofetil; Fecal Calprotectin
MeSH Terms: conditions — Diarrhea | interventions — Octreotide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diarrhea on MMF: Solid organ transplant recipients on MMF who develop diarrhea while taking the drug. Fecal calprotectin will be measured in their stool and Octreotide Acetate will be used to treat their diarrhea.
  Interventions: Drug: Octreotide Acetate

INTERVENTIONS:
Drug: Octreotide Acetate — Octreotide 100mcg SC q12h for 5 days

SUMMARY:
Prospective, observational pilot study of ten post-transplant patients presenting with diarrhea while taking Mycophenolate Mofetil (MMF). These patients will undergo a standard workup to confirm MMF induced diarrhea. A stool fecal calprotectin will be measured to determine if it may be helpful in confirming the diagnosis of MMF associated diarrhea. Once the diagnosis is confirmed, the patients will then be treated with a short course of subcutaneous Octreotide which has been shown to cure this type of diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between the ages of 18 and 75 years old who are solid organ transplant recipients followed at Toronto General Hospital on MMF referred to gastroenterology for diarrhea.

Exclusion Criteria:

1. Subjects with a known history of IBD or GVHD of the bowel.
2. Any subject receiving Octreotide for another indication.
3. Any patient unable to undergo endoscopy.
4. Any patient with a contraindication to Octreotide therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females between the ages of 18 and 75 years who are solid organ transplant recipients on mycophenolate mofetil (MMF) referred to gastroenterology at Toronto General Hospital for diarrhea.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Measurement of Fecal Calprotectin levels patients with diarrhea on MMF | 3 months

SECONDARY OUTCOMES:
Treatment of patients with MMF induced diarrhea with Octreotide | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maes B, Hadaya K, de Moor B, Cambier P, Peeters P, de Meester J, Donck J, Sennesael J, Squifflet JP. Severe diarrhea in renal transplant patients: results of the DIDACT study. Am J Transplant. 2006 Jun;6(6):1466-72. doi: 10.1111/j.1600-6143.2006.01320.x. PMID 16686772
- [Background] Allison AC, Eugui EM. Mycophenolate mofetil and its mechanisms of action. Immunopharmacology. 2000 May;47(2-3):85-118. doi: 10.1016/s0162-3109(00)00188-0. PMID 10878285
- [Background] Knoll GA, MacDonald I, Khan A, Van Walraven C. Mycophenolate mofetil dose reduction and the risk of acute rejection after renal transplantation. J Am Soc Nephrol. 2003 Sep;14(9):2381-6. doi: 10.1097/01.asn.0000079616.71891.f5. PMID 12937317
- [Background] Arns W. Noninfectious gastrointestinal (GI) complications of mycophenolic acid therapy: a consequence of local GI toxicity? Transplant Proc. 2007 Jan-Feb;39(1):88-93. doi: 10.1016/j.transproceed.2006.10.189. PMID 17275481
- [Background] Feichtiger H, Wieland E, Armstrong VW, Shipkova M. The acyl glucuronide metabolite of mycophenolic acid induces tubulin polymerization in vitro. Clin Biochem. 2010 Jan;43(1-2):208-13. doi: 10.1016/j.clinbiochem.2009.08.023. Epub 2009 Sep 8. PMID 19744471
- [Background] Calmet FH, Yarur AJ, Pukazhendhi G, Ahmad J, Bhamidimarri KR. Endoscopic and histological features of mycophenolate mofetil colitis in patients after solid organ transplantation. Ann Gastroenterol. 2015 Jul-Sep;28(3):366-373. PMID 26126799
- [Background] Liapis G, Boletis J, Skalioti C, Bamias G, Tsimaratou K, Patsouris E, Delladetsima I. Histological spectrum of mycophenolate mofetil-related colitis: association with apoptosis. Histopathology. 2013 Nov;63(5):649-58. doi: 10.1111/his.12222. Epub 2013 Sep 11. PMID 24025088
- [Background] Sydora MJ, Sydora BC, Fedorak RN. Validation of a point-of-care desk top device to quantitate fecal calprotectin and distinguish inflammatory bowel disease from irritable bowel syndrome. J Crohns Colitis. 2012 Mar;6(2):207-14. doi: 10.1016/j.crohns.2011.08.008. Epub 2011 Sep 7. PMID 22325175
- [Background] Ferreiro-Iglesias R, Barreiro-de Acosta M, Lorenzo-Gonzalez A, Dominguez-Munoz JE. Usefulness of a rapid faecal calprotectin test to predict relapse in Crohn's disease patients on maintenance treatment with adalimumab. Scand J Gastroenterol. 2016;51(4):442-7. doi: 10.3109/00365521.2015.1115546. Epub 2015 Nov 23. PMID 26595391
- [Background] Lorenz F, Marklund S, Werner M, Palmqvist R, Wahlin BE, Wahlin A. Fecal calprotectin as a biomarker of intestinal graft versus host disease after allogeneic hematopoietic stem cell transplantation. Sci Rep. 2015 Jan 21;5:7920. doi: 10.1038/srep07920. PMID 25605402
- [Background] Konikoff MR, Denson LA. Role of fecal calprotectin as a biomarker of intestinal inflammation in inflammatory bowel disease. Inflamm Bowel Dis. 2006 Jun;12(6):524-34. doi: 10.1097/00054725-200606000-00013. PMID 16775498